CLINICAL TRIAL: NCT07044973
Title: Dual-Target MR-guided Focused Ultrasound for Parkinson Disease
Brief Title: VIM+PTT MRgFUS for PD
Acronym: Dual-TargetFUS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Longsheng Pan, Professor, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 301-PD
Record Dates: First submitted 2025-06-23; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; VIM; PTT; MRgFUS
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ExAblate Treatment (Experimental): Participants will undergo a VIM and PTT thalamotomy using MRgFUS
  Interventions: Procedure: Transcranial focused ultrasound thalamotomy

INTERVENTIONS:
Procedure: Transcranial focused ultrasound thalamotomy — Thalamotomy Using Exblate

SUMMARY:
The objective of this prospective, single-arm, open-label study is to assess the safety and efficacy of the staged, dual-target（VIM+PTT thalamotomy）to treat Patiensts with Parkinson Disease using transcranial magnetic resonance guided focused ultrasound system ExAblate 4000, InSightec Ltd.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women age 30 years or older
2. Subjects who are able and willing to give informed consent and able to attend all study visits
3. Subjects with a diagnosis of idiopathic PD by UK Brain Bank Criteria as confirmed by a movement disorder neurologist at the site
4. Levodopa responsive as defined by at least a 30% reduction in MDS-UPDRS motor sub-scale in the ON vs OFF medication state
5. Disabling motor clinical features not optimally controlled by an adequate medication prescription. An adequate medication prescription is defined as a therapeutic dose of each medication or the development of side effects as the medication dose is titrated
6. Predominant disability from one side of the body (i.e unilateral or markedly asymmetric disease) as determined by movement disorders neurologist and neurosurgeon
7. Subjects should be on a stable dose of all PD medications for 30 days prior to study entry
8. Subjects are able to communicate sensations during the Exablate Transcranial procedure.
9. The thalamus must be apparent on MRI such that targeting of the Vim nucleus can be performed indirectly by measurement from a line connecting the anterior and posterior commissures of the brain.
10. Topographic coordinates of the pallidothalamic tract are localizable on Magnetic resonance imaging (MRI) so that it can be targeted by the ExAblate device.
11. Subject should have a Screening motor assessment of ≥ 30 while OFF medications on the MDS-UPDRS
12. Subject has a baseline CRST Part A score of 2 or above for postural or intention tremor severity in the upper extremity for the contralateral tremor side while on stable medication
13. Subject has a baseline CRST Part C score of 2 or above in any one of the items (speaking, eating, drinking, hygiene, dressing, writing, working, and social activities).

Exclusion Criteria:

1. Hoehn and Yahr stage in the ON medication state of 2 or lower
2. Presence of severe dyskinesia as noted by a score of 3 or 4 on questions 4.1 and 4.2 of the MDS-UPDRS
3. Presence of other central neurodegenerative disease suspected on neurological examination. These include: multisystem atrophy, progressive supranuclear palsy, corticobasal syndrome, dementia with Lewy bodies, and Alzheimer's disease
4. Any suspicion that Parkinsonian symptoms are a side effect from neuroleptic medications
5. Subjects who have had deep brain stimulation or a prior stereotactic ablation of the basal ganglia
6. Presence of significant cognitive impairment defined as score ≤ 21 on the Montreal Cognitive Assessment (MoCA) or presence of significant cognitive impairment as determined with a score ≤ 24 on the Mini Mental Status Examination (MMSE)
7. Unstable psychiatric disease, defined as active uncontrolled depressive symptoms, psychosis, delusions, hallucinations, or suicidal ideation. Subjects with stable, chronic anxiety or depressive disorders may be included provided their medications have been stable for at least 60 days prior to study entry and if deemed appropriately managed by the site neuropsychologist
8. Subjects with significant depression as determined following a comprehensive assessment by a neuropsychologist. Significant depression is being defined quantitatively as a score of greater than 14 on the Beck Depression Inventory
9. Legal incapacity or limited legal capacity as determined by the neuropsychologist
10. Subjects with unstable cardiac status including:

1. Unstable angina pectoris on medication 2. Subjects with documented myocardial infarction within six months of protocol entry 3. Significant congestive heart failure defined with ejection fraction < 40 4. Subjects with unstable ventricular arrhythmias 5. Subjects with atrial arrhythmias that are not rate-controlled 11. Severe hypertension (diastolic BP > 100 on medication) 12. History of or current medical condition resulting in abnormal bleeding and/or coagulopathy 13. Receiving anticoagulant (e.g. warfarin) or antiplatelet (e.g. aspirin) therapy within one week of focused ultrasound procedure or drugs known to increase risk or hemorrhage (e.g. Avastin) within one month of focused ultrasound procedure 14. Subjects with risk factors for intraoperative or postoperative bleeding as indicated by: platelet count less than 100,000 per cubic millimeter, a documented clinical coagulopathy, or INR coagulation studies exceeding the institution's laboratory standard 15. Patient with severely impaired renal function with estimated glomerular filtration rate <30 mL/min/1.73m2 (or per local standards should that be more restrictive) and/or who is on dialysis 16. Subjects with standard contraindications for MR imaging such as non-MRI compatible implanted metallic devices including cardiac pacemakers, size limitations, etc.

17. Significant claustrophobia that cannot be managed with mild medication 18. Subjects who weigh more than the upper weight limit of the MR table and who cannot fit into the MR scanner 19. Subjects who are not able or willing to tolerate the required prolonged stationary supine position during treatment 20. History of intracranial hemorrhage 21. History of multiple strokes, or a stroke within past 6 months 22. Subjects with a history of seizures within the past year 23. Subjects with brain tumors 24. Subjects with intracranial aneurysms requiring treatment or arterial venous malformations (AVMs) requiring treatment 25. Are participating or have participated in another clinical trial in the last 30 days 26. Any illness that in the investigator's opinion preclude participation in this study 27. Subjects unable to communicate with the investigator and staff 28. Pregnancy or lactation 29. Subjects with remarkable atrophy and poor healing capacity of the scalp (> 30% of the skull area traversed by the sonication pathway) will be excluded from this study 30. Subjects who have an overall Skull Density Ration lower than 0.30 as calculated from the screening CT

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Device and Procedure Related Adverse Events | 2 Years post treatment
  The cumulative sum of adverse events was followed through Year 2 of the study

SECONDARY OUTCOMES:
Clinical Rating Scale for Tremor (CRST) | Baseline,1 Month, 3 Months, 6 Months, 12 Months, 2 Years post treatment
  Sum of baseline and follow-up in upper extremity Tremor-Motor scores for the treated side is a sub-scale of Clinical Rating Scale for Tremor (CRST) Part A and Part B sum that was used to measure treated-side upper extremity tremor changes over time. Tremor-motor scores range from 0-32 points. Individual subject's scores at Baseline and Follow Up were calculated at baseline and follow-up visits averaged across subjects. Low scores are better (show improvement).
MDS-UPDRS (Movement Disorder Scale-Unified Parkinson's Disease Rating Scale), Part III | Baseline,1 Month, 3 Months, 6 Months, 12 Months, 2 Years post treatment
  MDS-UPDRS III is a scale that assesses all the motor features of PD (akinesia, tremor, rigidity, gait disturbance). Score range between 0 (no presence of motor features) and 132 (maximum score for all items).
Quality of life assessment with PDQ-39 | Baseline,1 Month, 3 Months, 6 Months, 12 Months, 2 Years post treatment
  Quality of life assessment with PDQ-39 (Range 0-156, scores are combined, the higher the score, the greater the level of clinical expression of Parkinson Disease, the worse clinical outcome is)

CONTACTS AND LOCATIONS:
Overall Officials: Longsheng Pan Professor, MD, Study Director — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China